CLINICAL TRIAL: NCT05940727
Title: Macroalgae Consumption - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Institute of Marine Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 332865
Record Dates: First submitted 2023-03-06; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Iodine Toxicity
Keywords: macroalgae; iodine; consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual macroalgae consumption (Active Comparator): Crossover design with habitual macroalgae consumption at baseline
  Interventions: Other: Habitual macroalgae consumption; Other: No macroalgae consumption
- Cessation of macroalgae consumption (Experimental): Cessation of macroalgae consumption as an experimental intervention.
  Interventions: Other: Habitual macroalgae consumption; Other: No macroalgae consumption

INTERVENTIONS:
Other: Habitual macroalgae consumption — The participant have a habitual macroalgae consumption at baseline.
Other: No macroalgae consumption — The participants exclude any macroalgae products from their diet

SUMMARY:
In this study, the aim is to investigate the food safety of macroalgae. There will be an analysis of macroalgae products for the concentration of cadmium, inorganic arsenic, and iodine in macroalgae, as well as measure the status of these elements in consumers. An investigation of the thyroid function of macroalgae consumers and the use of metabolomics to explore which biological changes occur when consuming seaweed and kelp and when the consumer excludes macroalgae from their diet will be performed.

DETAILED DESCRIPTION:
A group of consumers of macroalgae will be recruited to investigate their macroalgae intake and iodine, cadmium, and inorganic arsenic status and thyroid function. Iodine, cadmium, and inorganic arsenic have been selected since these elements have been described as relatively high in a previously published report from Norway. The goal is to recruit consumers of brown algae - especially kelp, and certain types of red algae, as these were the species with the highest content of iodine, cadmium, and arsenic, described in a previous publication. The participants will be asked to abstain from macroalgae for 6 weeks and again examine iodine status, cadmium and arsenic exposure, and thyroid function after the cessation period. A withdrawal period of 6 weeks has been chosen on the basis that it is calculated 6-8 weeks after Levaxin treatment for hypothyroidism before a new equilibrium can be expected and the effect of treatment on TSH can be assessed.

This study will provide new insight into the status of iodine, cadmium, and inorganic arsenic that macroalgae consumers have in urine and thyroid function after regular macroalgae consumption and after cessation of macroalgae intake. In addition, the study will provide descriptive data on macroalgae consumption, how it is eaten, how often, and how much. This can provide critical knowledge to the national and European authorities for food safety and public health advisers to evaluate the food safety of macroalgae.

ELIGIBILITY:
Inclusion Criteria:

* adults
* weekly consumer of macroalgae

Exclusion Criteria:

* pregnant
* known disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Consumption of macroalgae products | Through study completion, on average 6 weeks
  Assess the dietary consumption of macroalgae in consumers in the Bergen and Oslo area by 24hr recall and food frequency questionnaire
Levels of iodine, cadmium and inorganic arsenic in macroalgae products | Through study completion, on average 6 weeks
  Analyse the levels of iodine, cadmium and inorganic arsenic in macroalgae products used by the participants

SECONDARY OUTCOMES:
Levels of iodine | 6 weeks
  Analyse the levels of iodine in urine after intervention/usual macroalgae consumption
Levels of cadmium in urine | 6 weeks
  Analyse the levels of cadmium urine after intervention/usual macroalgae consumption
Levels of inorganic arsenic in urine | 6 weeks
  Analyse the levels of inorganic arsenic in urine after intervention/usual macroalgae consumption
Levels of creatinine in urine | 6 weeks
  Analyse the of creatinine in urine after intervention/usual macroalgae consumption
Thyroid function measure by thyroid-stimulating hormon | 6 weeks
  Measurement of thyroid-stimulating hormon (TSH) in serum after intervention/usual macroalgae consumption
Thyroid function measure by ree-triiodinetyronin | 6 weeks
  Measurement of free-triiodinetyronin (fT3) in serum after intervention/usual macroalgae consumption
Thyroid function measure by free thyroxine | 6 weeks
  Measurement of free thyroxine (fT4) in serum after intervention/usual macroalgae consumption
Thyroid function measure by Thyroid peroxidase antibody | 6 weeks
  Measurement of Thyroid peroxidase antibody (TPOAb) in serum after intervention/usual macroalgae consumption
Thyroid function measured by thyroglobulin | 6 weeks
  Measurement of thyroglobulin (Tg) in serum after intervention/usual macroalgae consumption
Thyroid function | 6 weeks
  Measurement of thyroid-stimulating hormon (TSH), free-triiodinetyronin (fT3), free thyroxine (fT4), Thyroid peroxidase antibody (TPOAb), thyroglobulin (Tg) in serum after intervention/usual macroalgae consumption
Metabolic changes | 6 weeks
  Measurement of metabolic changes by non-targeted metabolomics after intervention/usual macroalage consumption

CONTACTS AND LOCATIONS:
Overall Officials: Inger Aakre, PhD, Principal Investigator — Institute of Marine Research
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No